CLINICAL TRIAL: NCT05192395
Title: A Crossover, Randomized, Open-label, Comparison Study Between DWJ1525 and the Concomitant Use of DWP16001 and DWC202101 to Evaluate the Safety and Pharmacokinetic Properties in Healthy Volunteers
Brief Title: A Crossover Study of DWJ1525 to Evaluate the Safety and Pharmacokinetic Properties in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DW_DWJ1525101
Record Dates: First submitted 2022-01-05; First posted 2022-01-14 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2021-11

CONDITIONS: Healthy
MeSH Terms: interventions — Enavogliflozin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): fed state: period 1) DWJ15251, period 2) DWP16001 and DWC2021011 fased state: period 3) DWJ15251, period 4) DWP16001 and DWC2021011
  Interventions: Drug: DWJ1525; Drug: DWP16001; Drug: DWC202101
- Group B (Experimental): fed state: period 1) DWP16001 and DWC2021011, period 2) DWJ15251 fased state: period 3) DWP16001 and DWC2021011, period 4) DWJ15251
  Interventions: Drug: DWJ1525; Drug: DWP16001; Drug: DWC202101

INTERVENTIONS:
Drug: DWJ1525 — DWJ1525
Drug: DWP16001 — DWP16001
Drug: DWC202101 — DWC202101

SUMMARY:
A Randomized, Open-label, Single Oral Dosing, Two-sequence, and Four-period Crossover Study to Evaluate the Pharmacokinetics and Safety Between the Administration of DWJ1525 and the Co-administration of DWP16001 and DWC202101 for Healthy Subjects in Fed and Fasted State

DETAILED DESCRIPTION:
A single dose of the test (T) and two of the reference (R) products will be administered to the study subjects, according to a randomized, open-label, single oral dosing, two-sequence, and four-period crossover for healthy subjects in fed and fasted state study design.

A wash-out interval of at least 7 days will elapse between the each administrations.

The three investigational products will be administered with 150 mL of still mineral water on day 1 of the four study periods.

ELIGIBILITY:
Inclusion Criteria:

1. Before participating in the clinical trial, a person who fully explained the purpose, content, and characteristics of the clinical trial drug and signed a written consent form approved by the IRB of Bundang Cha Hospital to participate in this study according to his free will.
2. Healthy adults aged 19 or older at the time of screening.
3. Those who weigh more than 50 kg in men, weigh more than 45 kg in women, and have a body mass index (BMI) of 18.0 kg/m2 or more and less than 30.0 kg/m2 or less in women.

   * Body mass index (BMI) = Weight (kg) / [Height (m)] 2.

Exclusion Criteria:

1. A person with a clinically significant history in liver, kidney, digestive system, respiratory system, musculoskeletal system, endocrine system, neuropsychiatric system, blood and tumor system, cardiovascular system (including orthostatic hypotension), etc.
2. A history of gastrointestinal diseases (e.g., esophageal diseases such as Crohn's disease, esophageal achalasia, or esophageal stenosis) or surgery (except appendectomy, hernia, endoscopic polyp surgery, hemorrhoids, hemorrhoids, hemorrhoids, and healing surgery).
3. Those who are hypersensitive to other drugs (aspirin, antibiotics, etc.) or have a history of clinically significant hypersensitivity reactions, including clinical drug ingredients (Enavogliflozin, Metformin) and homogeneous (SGLT2 inhibitors)
4. A person who shows the following results in the inspection items conducted during screening.

   * Blood ALT, AST, Total bilirubin > twice the upper limit of the normal range
   * The glomerular filtration rate (e-GFR) <90 mL/min/1.73 m2 (using the CKD-EPI method)
   * If the blood glucose level is greater than 125 mg/dL or less than 60 mg/dL,
   * After more than 3 minutes of rest, systolic blood pressure > 150 mmHg or <90 mmHg, or diastolic blood pressure > 100 mmHg or <50 mmHg in vital signs measured at the seat.
5. A person whose abnormal results were judged to be clinically significant in screening test items (examination, vital signs, electrocardiogram, physical examination, blood, urinary examination, etc.) other than those mentioned in paragraph 4).
6. Drugs that do not affect the safety and research results of the subject may be available within 14 days of the first administration of clinical trial drugs (including herbal medicines), general medicines (including vitamins), and health functional foods.)
7. Those who took other clinical trial drugs within 180 days before the first scheduled date of administration of clinical trial drugs (however, the criteria for termination of participation in previous clinical trials are calculated as one day based on the last administration date.)
8. A person who has continuously consumed more than 21 units/week (1 unit = 10g = 12.5 mL) within 6 months of screening or cannot abstain from drinking alcohol from 3 days before the first administration of clinical trial drugs to the last visit.

   ☞ Alcohol amount (g) = Consumption (mL) x frequency (%) x 0.8
9. Those who smoke more than 10 cigarettes a day within 6 months of screening and who cannot quit smoking excessively from 3 days before the first clinical trial drug administration to the last visit or quit smoking from the date of hospitalization to the last blood collection.
10. A person who donated whole blood within 8 weeks before the first scheduled date of administration of clinical trial drugs, or who donated whole blood within 4 weeks (plasma, platelet), or did not agree to prohibit blood donation until 30 days after the last administration date.
11. Those who did not agree to stop taking diet (e.g., grapefruit) that could affect the absorption, distribution, metabolism, and excretion of drugs from three days before the first administration of clinical trial drugs to the last blood collection.
12. Those who do not agree to consume excessive caffeine (400 mg/day) from 3 days before the first clinical trial drug administration to the last visit or to stop consuming caffeine-containing foods from the date of hospitalization to the time of blood collection.
13. A person who does not use the appropriate contraceptive method recognized by his/her spouse or partner from the time of written consent to the subject until two weeks after the date of administration of the last clinical trial drug.
14. Pregnant women or lactating women identified during screening.
15. Other persons who have judged that they are inappropriate to participate in this examination as judged by the tester.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2022-04-15 (Actual); Primary Completion 2022-05-24 (Actual); Study Completion 2022-05-24 (Actual)

PRIMARY OUTCOMES:
AUClast | At pre-dose (0) and 0.25 to 72 hours post dose
  AUClast of plasma DWP16001 and DWC202101
Cmax | At pre-dose (0) and 0.25 to 72 hours post dose
  Cmax of plasma DWP16001 and DWC202101

CONTACTS AND LOCATIONS:
Locations (1):
- CHA unuversity bundang medical center, Seongnam, South Korea